CLINICAL TRIAL: NCT02363465
Title: Echographic Measurement of Skin Thickness at the Deltoid and Proximal Forearm in Adults
Brief Title: Echographic Measurement of Skin Thickness
Status: Completed | Type: Observational
Sponsor: Novosanis NV (Industry)
Responsible Party: Sponsor
Other Study IDs: 300201523257
Record Dates: First submitted 2015-02-04; First posted 2015-02-16 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Skin Thickness
Keywords: skin thickness; high-frequency ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Participants aged 18-30 years: Echographic measurement of skin thickness at the proximal forearm and the deltoid region in participants aged 18-30 years.
  aimed number: 12 male & 12 female maximum number: 15 male & 15 female
  Interventions: Other: Echographic measurement of skin thickness
- Participants aged 31-40 years: Echographic measurement of skin thickness at the proximal forearm and the deltoid region in participants aged 31-40 years.
  aimed number: 12 male & 12 female maximum number: 15 male & 15 female
  Interventions: Other: Echographic measurement of skin thickness
- Participants aged 41-50 years: Echographic measurement of skin thickness at the proximal forearm and the deltoid region in participants aged 41-50 years.
  aimed number: 12 male & 12 female maximum number: 15 male & 15 female
  Interventions: Other: Echographic measurement of skin thickness
- Participants aged 51-65 years: Echographic measurement of skin thickness at the proximal forearm and the deltoid region in participants aged 51-65 years.
  aimed number: 12 male & 12 female maximum number: 15 male & 15 female
  Interventions: Other: Echographic measurement of skin thickness

INTERVENTIONS:
Other: Echographic measurement of skin thickness — (Epi)Dermal thickness at the proximal forearm and the deltoid region will be measured using imaging technology, more specifically high-frequency ultrasound (20-40 MHz) in B-mode (VEVO 2100®, Visual Sonics). This non-invasive measuring technique has already been proven to be accurate.
  The echographic measurement will be performed on the left and right deltoid region and on two sides of the proximal forearm. Both the dorsal part and the volar/palmar part of the proximal forearm will be investigated. Ultrasound will be executed using gel (Aquasonic®) to optimize imaging.

SUMMARY:
To optimize a medical device for intradermal injection, knowledge concerning the thickness of epidermis and dermis at the proximal forearm is required. Since scientific knowledge is lacking, the investigators will examine the skin thickness (epidermis and dermis) of adults using imaging technology (High Frequency Ultrasound). The investigators hypothesize that they are able to correlate the thickness of the (epi)dermis to a specific combination of parameters age, gender, and BMI.

Based on these results, the investigators can define which needle type and length is needed to correctly perform injections into the dermal layer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Age: 18-65 years
* Dutch-speaking
* Caucasian

Exclusion Criteria:

* Pregnancy or lactating
* Using ointment, crème, or gels based on corticoids
* Suffering from skin diseases (psoriasis, burning wounds)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited in the vicinity of the university and its university hospital of Antwerp, in the period of January 2015 until April 2015.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
skin thickness (in milimeters) of the proximal forearm dorsal (both left and right) | 10 minutes
skin thickness (in milimeters) of the proximal forearm ventral (both left and right) | 10 minutes
skin thickness (in milimeters) of the deltoid region (both left and right) | 10 minutes

SECONDARY OUTCOMES:
Body Mass Index | at the moment of entering the study
Age | at the moment of entering the study
sex | at the moment of entering the study

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Vankerckhoven, PhD, Principal Investigator — CEO
Locations (1):
- Department of Pharmaceutical Sciences; Laboratory of Physiopharmacology; University of Antwerp; Campus Drie Eiken, Wilrijk, Antwerp, Belgium

REFERENCES:
- [Derived] Van Mulder TJ, de Koeijer M, Theeten H, Willems D, Van Damme P, Demolder M, De Meyer G, Beyers KC, Vankerckhoven V. High frequency ultrasound to assess skin thickness in healthy adults. Vaccine. 2017 Mar 27;35(14):1810-1815. doi: 10.1016/j.vaccine.2016.07.039. Epub 2016 Aug 3. PMID 27496276